CLINICAL TRIAL: NCT06675747
Title: Ultrasonographic Evaluation of the Effect of Occlusal Splint Therapy on the Masseter and Temporal Muscles in Patients with Myofascial Pain Syndrome
Brief Title: Evaluation of the Effect of Occlusal Splint Use on Masticatory Muscles
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Berk Bilgen, PhD DDS, Research Assistant at Department of Prosthodontics, Istanbul University
Other Study IDs: 2024/03-Rev-1
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Myofascial Pain - Dysfunction Syndrome of TMJ
Keywords: myofascial pain; temporomandibular disorders; occlusal splint; ultrasonography; masseter muscle; temporal muscle
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: Female patients will be selected from those who present with various maxillofacial muscle pain complaints to the 'Temporomandibular Disorders Clinic' at the Department of Prosthodontics, Istanbul University Faculty of Dentistry. Female patients diagnosed with myofascial pain syndrome and for whom occlusal splint therapy is planned will be included in the study will be selected from this patient group.
  Interventions: Other: Ultrasound imaging

INTERVENTIONS:
Other: Ultrasound imaging — To investigate the mechanism of action of occlusal splints, a routinely applied treatment method for myogenic temporomandibular disorders, ultrasound images will be taken from all patients before and after treatment, and measurements will be conducted based on these images.

SUMMARY:
"Female patients who applied to the 'Temporomandibular Disorders (TMD) Clinic' at the Department of Prosthodontics, Istanbul University Faculty of Dentistry, with complaints of muscle pain in the maxillofacial region and who are diagnosed with myofascial pain syndrome based on the results of their examination and the Temporomandibular Disorders Diagnostic Criteria (TMD-DC) form they completed, will be included in the study. Occlusal splint therapy will be initiated for these patients. Before starting occlusal splint therapy, ultrasound images will be taken from the patients. Subsequently, the patients will undergo routine occlusal splint therapy without any intervention in their 12-week treatment process. At the end of the 12-week treatment protocol, during the final control session, patients will fill the TMD-DC form again, and the two forms will be compared to evaluate changes in their clinical symptoms and pain. Additionally, a second ultrasound imaging will be taken during the same session. In this imaging, the thickness and blood flow of the masseter and temporal muscles will be examined, and comparisons will be made with the pre-treatment ultrasound. In this way, the effects of occlusal splints on muscle morphology and blood flow will be evaluated."

DETAILED DESCRIPTION:
The study is designed as a prospective observational clinical study. Female patients will be selected from those who applied to the 'Temporomandibular Disorders (TMD) Clinic' at the Department of Prosthodontics, Istanbul University Faculty of Dentistry with various maxillofacial muscle pain complaints. Only female patients will be included in the study, as temporomandibular disorders caused by masticatory muscles are observed approximately four times more frequently in women than in men, and for muscle studies, it is recommended to examine a single gender group for scientific consistency. (Studies combining male and female participants have been found to have lower reliability due to significant differences in muscle volume and thickness between genders.)

During the examination of these patients, Temporomandibular Disorders Diagnostic Criteria (TMD-DC) forms will be completed to reach an accurate diagnosis. Female patients diagnosed with myofascial pain syndrome and for whom occlusal splint therapy is planned will be included in the study. Individuals participating in the study will be selected from this patient group. Before starting occlusal splint therapy, ultrasound (USG) images will be taken, focusing on the masseter muscle, temporal muscle, facial artery, maxillary artery, temporal artery, and external carotid artery.

The 12-week routine treatment of these patients will proceed without any intervention. At the end of their treatment, when patients return for their final control session, they will complete the TMD-DC forms again to evaluate changes in symptoms and pain. (Evaluations will be made based on Jaw Functional Limitation Scale (JFLS) scores, pain rating, maximum mouth opening, pain during palpation of the masseter muscle, and pain during palpation of the temporal muscle.)

During the same session, a second USG will also be taken. The results obtained will be compared with the initial USG images taken before treatment. In these images, the thickness, length, and elastography values of the masseter and temporal muscles, both at rest and during clenching, will be measured, and the blood flow rates in the arteries will be assessed. Arterial assessment will be based on (Pulsatility Index) PI, (Resistive Index) RI, Peak Systolic Velocity (PS), End Diastolic Velocity (ED) , and Time-averaged maximum speed (TAMAX) values. Thus, the effect of occlusal splint therapy on muscle morphology and blood flow will be evaluated."**

ELIGIBILITY:
Inclusion Criteria:

* Female patients who presented with muscle pain complaints to Istanbul University Faculty of Dentistry
* Patients diagnosed with myospasm and/or myofascial pain syndrome in the masseter and/or temporal muscles
* Patients who have not previously received occlusal splint therapy
* Patients without any physical or mental disabilities
* Patients over the age of 18
* Patients with no missing teeth

Exclusion Criteria:

* Patients with any temporomandibular disorders (TMD) other than masticatory muscle disorders
* Male patients
* Patients who have previously received any TMD treatment
* Patients under the age of 18
* Patients with any physical or mental disabilities
* Patients with missing teeth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females were eligible to participate
Study Population: Female patients will be selected from those who present with various maxillofacial muscle pain complaints to the 'Temporomandibular Disorders Clinic' at the Department of Prosthodontics, Istanbul University Faculty of Dentistry. Only female patients will be included in the study, as temporomandibular disorders caused by masticatory muscles are observed approximately four times more frequently in women than in men, and for muscle studies, it is recommended to examine a single gender group for scientific consistency. (Studies combining male and female participants have been found to have lower reliability due to significant differences in muscle volume and thickness between genders.) Female patients diagnosed with myofascial pain syndrome and for whom occlusal splint therapy is planned will be included in the study.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
"Changes observed after treatment in the temporal and masseter muscles, as well as in the blood flow of their associated arteries." | 12 weeks
  Ultrasound images taken before and after the application of the occlusal splint will be compared to assess the length, elastography, thickness in the open-mouth position, and thickness during clenching of the masseter and temporal muscles. This comparison will determine the effect of occlusal splints on these two muscles. Additionally, blood flow in the facial artery, temporal artery, maxillary artery, and external carotid artery will be examined to evaluate whether the treatment causes any changes in arterial blood flow.

SECONDARY OUTCOMES:
The effect of occlusal splints on clinical symptoms | 12 weeks
  The effect of the occlusal splint on reducing the patient's muscle pain levels, jaw opening capacity, Jaw Functional Limitation Score (JFLS), and pain levels during palpation of the relevant muscles will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Olcay Sakar, Prof. Dr. Lecturer, Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yalcin ED, Aslan Ozturk EM. Ultrasonographic evaluation of the effect of splint therapy on masseter muscle and blood flow in patients with bruxism. Cranio. 2025 Jan;43(1):135-143. doi: 10.1080/08869634.2022.2088575. Epub 2022 Jul 11. PMID 35816105